CLINICAL TRIAL: NCT01094028
Title: Intraumbilical Vein Injection of Oxytocin in Routine Practice for Active Management of the Third Stage of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: No sponsor, No sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07
Record Dates: First submitted 2010-03-22; First posted 2010-03-26 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2009-12

CONDITIONS: Labor
Keywords: Blood loss in the third and fourth stage of labor and the duration of third stage of labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saline group (Experimental): Only 30 mL of saline was injected directly in the umbilical vein after clamping. The injection was performed with a 30-mL syringe and an 18-gauge needle around 1 to 2 cm from the introitus. The solution was injected slowly over 1 minute and at the end of the injection, the solution was milked toward the cord insertion.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 20 IU of oxytocin diluted with 26 ml of saline.The medication was injected directly in the umbilical vein after clamping. The injection was performed with a 30-ml syringe and an 18-gauge needle around 1 to 2 cm from the introitus. The solution was injected slowly over 1 minute, and at the end of the injection, the solution was milked toward the cord insertion

SUMMARY:
During the first hours that follow the birth of the baby (third and fourth stages of labor), complications are common and can threaten the mother's life. The most common complication is postpartum hemorrhage (PPH), which remains a leading cause of maternal mortality (25.0%) especially in developing countries .Three to five percent of deliveries are complicated by PPH and is 50 times more common in developing countries. Retained placenta is an another complication of third stage of labor. It complicates 0.1-2 % of deliveries . Without prompt treatment, women are at high risk of hemorrhage. At present, treatment is by manual removal of placenta, which needs an operating theatre, a surgeon, and an anaesthetist-facilities that are often unavailable to women in resource-poor settings. As a result, this condition has a case fatality rate of nearly 10% in rural communities.

The length of the third stage of labor, and its subsequent complications depends on a combination of the length of time it takes for placental separation and the ability of the uterine muscle to contract. Principal management of the third stage of labor is aimed at reducing the time of delivery of placenta so minimising serious adverse effects, such as blood loss and retained placenta. Active management of the third stage of labor, which includes prophylactic injection of 10 units of oxytocin within two minutes of birth, early clamping of the umbilical cord and controlled cord traction (CCT), is recommended by WHO for PPH prevention .

Umbilical vein oxytocin injection directs the treatment to the placental bed and uterine wall, resulting in an earlier uterine contraction and placental separation. However, very limited published literature is available, which evaluated the effect of umbilical vein oxytocin injection in routine practices for active management of the third stage of labor. The purpose of this investigation was to find out the beneficial effect of adding intraumbilical vein oxytocin in reducing the blood loss during third and fourth stages of labor, length of third stage of labor, and reduction in the incidence of manual removal of retained placenta.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 37 and 42 weeks
* singleton pregnancy
* live fetus
* cephalic presentation
* neonatal birth weight of 2500-4500 g
* parity between one and five
* maternal age < 35 years
* vaginal birth

Exclusion Criteria:

* blood pressure ≥ 140/90mmHg
* placenta previa
* placental abruption
* a history of any bleeding during pregnancy
* a history of curettage
* cesarean section or any uterine scar
* a history of postpartum hemorrhage
* polyhydramnios
* signs or symptoms of maternal infection
* known uterine anomalies
* history of any drug use during labor
* abnormal placentation)
* coagulation defects
* instrumental deliveries
* hemoglobin concentration < 8 g/dL
* history of anticoagulant drugs
* beta-mimetic medications during pregnancy
* prolongation of the first stage of labor > 15 hours.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 412 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
the amount of blood loss in third and fourth stages of labor | The end of the delivery to 2 hours after birth.

SECONDARY OUTCOMES:
duration of the third stage
  The duration of the third stage of labor was defined as the time difference (in minutes) between delivery of the infant and delivery of the placenta. The time interval was measured by the nurse attending the delivery and confirmed by the physician using a digital stop clock. The clock was started as soon as baby's body was totally delivered and stopped as soon as the placenta was completely expulsed.

REFERENCES:
- [Derived] Gungorduk K, Asicioglu O, Besimoglu B, Gungorduk OC, Yildirm G, Ark C, Tekirdag AI. Using intraumbilical vein injection of oxytocin in routine practice with active management of the third stage of labor: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):619-624. doi: 10.1097/AOG.0b013e3181edac6b. PMID 20733444